CLINICAL TRIAL: NCT01496664
Title: Coronary Hybrid Revascularisation Study Registry on Treatment of Significant Coronary Artery Disease by Combined Bypass Operation (CABG) and Catheter Based Treatment (PCI)
Brief Title: Coronary Hybrid Revascularisation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, phd, Aarhus University Hospital Skejby
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-20100152
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Significant Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Result of combined CABG and PCI treatment (Experimental): The registry is to assess results of combined operative and catheter based (hybrid procedure) treatment of patients with significant coronary artery disease using essential clinical and angiographic parameters.
  Interventions: Procedure: Combined CABG and PCI

INTERVENTIONS:
Procedure: Combined CABG and PCI — Coronary artery bypass grafting Percutaneous coronary intervention

SUMMARY:
The purpose of the registry is to assess results of combined operative and catheter based (hybrid procedure) treatment of patients with significant coronary artery disease using essential clinical and angiographic parameters.

Based on existing literature we expect the results of coronary artery bypass grafting of the anterior descendent coronary artery (LAD), segment 1 and 2, using the so-called mammary artery graft, to be superior to stent treatment of the same artery.

At the same time a catheter based intervention using balloon, bare metal stents (BMS) or drug eluting stents (DES) seems to be a better treatment that a saphenous vein graft for other coronary arteries than the LAD. I.e. the right coronary artery (RCA) and the left circumflex coronary artery (CX).

Therefore, we expect a combination of the mentioned surgical and catheter based techniques to be a better treatment than bypass operation or catheter based intervention alone.

DETAILED DESCRIPTION:
A total of 150 consecutive patients will be included in the study. The patients will have a coronary artery narrowing located to the LAD, which can be treated with a mammary graft, and a stenosis located to other coronary arteries (RCA and CX), which can be treated by balloon or stent.

The patients included in the study will be recruited from patients who are referred to the Department of Cardiology/Department of Thoracic Surgery, Aarhus University Hospital, Skejby for treatment of significant coronary artery disease. We will not announce for patients, and the patients will not receive a honorarium for participation.

The first 100 patients will be treated i two seances; operation and stent treatment with few days interval. The last 50 patients will be treated in a hybrid operation room with operation and stent treatment in the same seance.

ELIGIBILITY:
Inclusion Criteria:

* Stable, unstable angina pectoris and ACS.
* Significant stenosis of LAD, segment 1 or 2 and of other coronary arteries.
* The patient can be treated with a mammary graft to LAD and by balloon or stent of other lesions.
* Signed informed consent must be available.

Exclusion Criteria:

* Earlier cardiac surgery
* Treatment with coronary stent within one year.
* ST-elevation infarction within 24 hours.
* Coronary artery lesions located to LAD, segment 1 or 2, which cannot be treated by coronary bypass operation.
* Stenosis of diagonal branches, CX artery and the right coronary artery, which cannot be treated by PCI.
* Expected survival <1 year following successful treatment.
* Allergy to aspirin, clopidogrel, ticlopidine and/or prasugrel.
* Allergy to sirolimus, everolimus, zotarolimus og biolimus

For the patients treated with coronary hybrid intervention in the same seance further exclusion criteria:

Known disorder of the bloods ability to coagulate (such as renal failure (dialysis or renal creatinine clearance < 50ml/min), congenital coagulopathy, needs for anticoagulant treatment before surgery) Previous gastrointestinal bleeding or previous cerebral

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of death, stroke, MI and new revascularisation (PCI or CABG) MACCE | After 1 year

SECONDARY OUTCOMES:
Combined endpoint of death, stroke, MI and new revascularisation. | After 1 month and after 1, 3 and 5 years
Individual endpoints of death, stroke, MI and new revascularisation. | After 1 month and after 1, 3 and 5 years
Death | Baseline, 1 month, 1, 2, 3, 4 and 10 years
Procedure related biomarker release | Baseline, 1, 3 and 5 year
Reoperation for bleeding | Baseline, 1, 3 and 5 year
Operation for suspected sternal infection | Baseline, 1, 3 and 5 year
CT verified pulmonary embolism | Baseline, 1, 3 and 5 year
CCS angina class | 1, 3 and 5 year
NYHA function class | 1, 3 and 5 year
Duration of hospitalisation related to the index treatment | Baseline
Duration of admission for the index treatment | Baseline
Angiographic endpoints | 1 year
  Presence of significant narrowing or occlusion of mammary or vein graft, or lesions treated with stent or balloon.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Rimestad JM, Christiansen EH, Modrau IS. One-year cost-effectiveness and safety of simultaneous hybrid coronary revascularization versus conventional coronary artery bypass grafting. Interact Cardiovasc Thorac Surg. 2019 Aug 1;29(2):217-223. doi: 10.1093/icvts/ivz083. Epub 2019 Mar 21. PMID 30903175
- [Derived] Modrau IS, Holm NR, Maeng M, Botker HE, Christiansen EH, Kristensen SD, Lassen JF, Thuesen L, Nielsen PH; Hybrid Coronary Revascularization Study Group. One-year clinical and angiographic results of hybrid coronary revascularization. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1181-6. doi: 10.1016/j.jtcvs.2015.08.072. Epub 2015 Aug 28. PMID 26432721
- [Derived] Modrau IS, Nielsen PH, Botker HE, Christiansen EH, Krusell LR, Kaltoft AK, Maeng M, Terkelsen CJ, Kristensen SD, Lassen JF, Thuesen L. Feasibility and early safety of hybrid coronary revascularisation combining off-pump coronary surgery through J-hemisternotomy with percutaneous coronary intervention. EuroIntervention. 2015 Feb;10(10):e1-6. doi: 10.4244/EIJV10I10A195. PMID 24103704
- See also: Feasibility and early safety of hybrid coronary revasculatisation combining off-pump coronary surgery through J-hemisternotomy with percutaneous coronary intervention — https://eurointervention.pcronline.com/article/feasibility-and-early-safety-of-hybrid-coronary-revascularisation-combining-off-pump-coronary-surgery-through-j-hemisternotomy-with-percutaneous-coronary-intervention
- See also: One year clinical and angiographic results of hybrid coronary revascularisation — https://www.ncbi.nlm.nih.gov/pubmed/26432721
- See also: Related Info — https://eurointervention.pcronline.com/article/feasibility-and-early-safety-of-hybrid-coronary-revascularisation-combining-off-pump-coronary-surgery-through-j-hemisternotomy-with-percutaneous-coronary-intervention